CLINICAL TRIAL: NCT02972554
Title: Beta-Blockers and Inflammatory Responses to Acute Psychosocial Stress
Brief Title: Does Propranolol Attenuate Inflammatory Responses to a Psychological Stressor?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16-2498
Record Dates: First submitted 2016-10-26; First posted 2016-11-23 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-01

CONDITIONS: Stress, Psychological; Inflammation; Cortisol; Sympathetic Nervous System
MeSH Terms: conditions — Stress, Psychological; Inflammation | interventions — Propranolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propanolol Hydrochloride (Experimental): This is the experimental group given the beta-blocker
  Interventions: Drug: Propanolol hydrochloride
- Placebo (Placebo Comparator): This is the control group given a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propanolol hydrochloride — One-time dose of 40mg of propranolol
  Other Names: Inderal
  Arms: Propanolol Hydrochloride
Other: Placebo — Outside casing matching that of active drug
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study of propranolol will shed important light on how sympathetic nervous system (SNS) activation influences psychological and inflammatory responses to acute stress. Results from this study will inform both the basic science literature that is attempting to map the physiological mechanisms by which psychological stress may lead to poor mental and physical health, and may also ultimately have therapeutic relevance for individuals who are experiencing high levels of stress that is putting their health at risk. Utilizing a psychopharmacological approach allows for the circumvention of many of the challenges of conducting this research in human populations, and will allow for conclusions regarding causality, given that SNS activation will be experimentally manipulated, rather than relying on correlational measures of SNS activity that are difficult to assess and are not appropriate for asking if SNS activity causes changes in psychology and biology.

DETAILED DESCRIPTION:
Psychological stress is implicated in the onset and progression of many common and costly chronic diseases, including cardiovascular disease, chronic pain conditions, and major depressive disorder (Cohen et al., 2007; Kendler et al., 1999; Steptoe and Kivimäki, 2012). An emerging body of evidence suggests that inflammation, indexed via levels of pro-inflammatory cytokines and reactive proteins, may be a key biological mechanism by which stress affects health (Baker et al., 2012; Miller et al., 2009; Slavich et al., 2010). Indeed, psychological stressors can induce increases in inflammation (Slavich and Irwin, 2014; Kiecolt-Glaser et al., 2003; Rohleder, 2014; Steptoe et al., 2007), and greater levels of inflammation may contribute to the development of disease (Capuron and Miller, 2004; Choy and Panayi, 2001; DellaGiola and Hannestad, 2010; Raison and Miller, 2013; The Emerging Risk Factors Collaboration, 2010). Despite this growing literature linking stress, inflammation, and poor health, little is known about the precise physiological mechanisms linking psychological stress and increases in inflammation.

One hypothesized mechanism that may translate psychological stress into increases in levels of inflammation is activation of the sympathetic nervous system (SNS). The SNS is part of the autonomic nervous system and is primarily indexed by release of the catecholamines epinephrine (adrenaline) and norepinephrine (noradrenaline). Prior research in non-human animal models has shown that stress-induced SNS activation leads to increases in levels of pro-inflammatory cytokines inflammation (Bierhaus et al., 2003; DeRijk et al., 1994; Kop et al., 2008; van Gool et al., 1990), while pharmacologically blocking sympathetic activation attenuates the inflammatory response to stress (Bierhaus et al., 2003). However, no known human studies to date have examined the relationship between psychological stress, SNS activation, and inflammation. The present study is designed to address this major gap in our knowledge of the physiological mechanisms that may link stress and disease.

A potential reason for the lack of human research linking stress, SNS activation, and inflammation is that SNS activity is difficult to measure. Indeed, adrenaline and noradrenaline are released into the bloodstream very rapidly during a stressor, making their kinetics difficult to capture during typical laboratory-based stress paradigms. Indirect measures of SNS activity may be acquired using psychophysiological approaches that involve peripheral measures of electrical activity and efficiency of the heart; however, these methods provide only indirect indicators of SNS activity, making them subject to criticism in the psychoneuroimmunology community.

To circumvent these issues with assessment of SNS activity, the present study will employ a psychopharmacological approach to experimentally block SNS activity using the drug propranolol. Propranolol is a beta-blocker medication that is very commonly prescribed by physicians in the United States for the treatment of hypertension, given that it blocked adrenergic receptors that lead to relaxation of the cardiac muscle and smooth muscle tissue. Interestingly, propranolol is also sometimes prescribed to individuals who have performance anxiety (i.e., public speaking anxiety), as reducing SNS activity (i.e., eliminating the increased heart rate, blood pressure, sweaty palms, etc., that typically accompany anxiety-provoking situations) has been anecdotally observed to decrease perceptions of stress during these situations. Psychological scientists have recently become more interested in the role SNS activity may play in the formation and reconsolidation of fear memories, and a number of studies have now used propranolol to investigate if blocking SNS activity may help treat individuals with Post-Traumatic Stress Disorder (PTSD; Pitman et al., 2002; Vaiva et al., 2003). However, only one known study to date has investigated if propranolol reduces stress-induced immune system activation (Benschop et al., 1994), and this (now dated) study did not specifically explore if propranolol reduces inflammatory responses to stress. Furthermore, no known studies have examined if blocking SNS activity with propranolol changes individuals' appraisals of the stressful situation, or their affective responses to stress. Results from this study will complement and extend the existing work on how SNS activity affects fear memories and stress by focusing on how propranolol affects inflammatory and psychological responses to a stressor.

In addition to these primary goals of the present study, the investigators will also explore the role of SNS activation in a number of additional exploratory tasks that are hypothesized to be affected by sympathetic arousal. More specifically, the investigators will examine if exposure to propranolol eliminates implicit biases toward out-group members (in this case, African Americans), given that a very large literature suggests that many White Americans hold implicit biases against African Americans (Wittenbrink et al., 1997; Nosek et al., 2002). While it has been hypothesized that sympathetic arousal based on cultural stereotypes associating African Americans with negativity may be leading to these implicit biases, no known studies have investigated this issue. The investigators will also explore of SNS activation is critical for empathy, or individual's ability to understand the emotional states of others, for avoiding risky decisions, and for moral judgments. Thus, this study will also answer a number of exploratory, unanswered questions in social psychology regarding the role that sympathetic arousal plays in some of our most fundamental psychological processes.

In sum, this randomized, double-blind, placebo-controlled study of propranolol will shed important light on how SNS activation influences our psychological and inflammatory responses to stress. Results from this study will inform both the basic science literature that is attempting to map the physiological mechanisms by which psychological stress may lead to poor mental and physical health, and may also ultimately have therapeutic relevance for individuals who are experiencing high levels of stress that is putting their health at risk. By utilizing psychopharmacological approaches, the investigators will circumvent many of the challenges of conducting this research in human populations. The investigators will also be in a place to draw strong conclusions regarding causality, given that they will have experimentally manipulated SNS activation, rather than relying on correlational measures of SNS activity that are difficult to assess and are not appropriate for asking if SNS activity causes changes in psychology and biology.

ELIGIBILITY:
Inclusionary Criteria:

1. Healthy volunteers
2. Age 18-25
3. Fluent in English

Exclusionary Criteria:

1. presence or history of chronic physical illness (especially disorders with an inflammatory component, such as rheumatoid arthritis, asthma, allergies, or issues that can affect the heart, including low-blood pressure or other heart conditions)
2. presence or history of psychiatric illness (depression, anxiety)
3. any current prescription medication use
4. currently pregnant or planning to become pregnant
5. engagement in a number of health--compromising behaviors that may affect levels of pro-inflammatory cytokines, including cigarette smoking, excessive caffeine intake and sleep disturbance (e.g., working night shifts)
6. body mass index (BMI) greater than 30, given that adiposity is known to relate to baseline levels of inflammation
7. anxiety about or previous history of problems with blood draws (e.g., fainting)
8. any reported heart conditions
9. history of fainting spells
10. low pulse, as measured at beginning of session I (below 60)
11. low blood pressure, as measured at beginning of session I (below 80)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keely A Muscatell, Ph.D, Principal Investigator — University of North Carolina at Chapel Hill, Psychology & Neuroscience
Locations (1):
- Howell Hall, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler N, Stewart J. The MacArthur Scale of Subjective Social Status. 2007. http://www.macses.ucsf.edu.
- [Background] Baker DG, Nievergelt CM, O'Connor DT. Biomarkers of PTSD: neuropeptides and immune signaling. Neuropharmacology. 2012 Feb;62(2):663-73. doi: 10.1016/j.neuropharm.2011.02.027. Epub 2011 Mar 22. PMID 21392516
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Barrett LF. Feelings or words? Understanding the content in self-report ratings of experienced emotion. J Pers Soc Psychol. 2004 Aug;87(2):266-81. doi: 10.1037/0022-3514.87.2.266. PMID 15301632
- [Background] Beck, A.T., Steer, R.A., & Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] Benschop RJ, Nieuwenhuis EE, Tromp EA, Godaert GL, Ballieux RE, van Doornen LJ. Effects of beta-adrenergic blockade on immunologic and cardiovascular changes induced by mental stress. Circulation. 1994 Feb;89(2):762-9. doi: 10.1161/01.cir.89.2.762. PMID 7508828
- [Background] Blascovich, J. & Mendes, W. B. (2000). Challenge and threat appraisals: The role of affective cues. In Forgas, J. (Ed.). Feeling and thinking: The role of affect in social cognition (pp. 59-82). New York, NY: Cambridge University Press.
- [Background] Bierhaus A, Wolf J, Andrassy M, Rohleder N, Humpert PM, Petrov D, Ferstl R, von Eynatten M, Wendt T, Rudofsky G, Joswig M, Morcos M, Schwaninger M, McEwen B, Kirschbaum C, Nawroth PP. A mechanism converting psychosocial stress into mononuclear cell activation. Proc Natl Acad Sci U S A. 2003 Feb 18;100(4):1920-5. doi: 10.1073/pnas.0438019100. Epub 2003 Feb 10. PMID 12578963
- [Background] Capuron L, Miller AH. Cytokines and psychopathology: lessons from interferon-alpha. Biol Psychiatry. 2004 Dec 1;56(11):819-24. doi: 10.1016/j.biopsych.2004.02.009. PMID 15576057
- [Background] Choy EH, Panayi GS. Cytokine pathways and joint inflammation in rheumatoid arthritis. N Engl J Med. 2001 Mar 22;344(12):907-16. doi: 10.1056/NEJM200103223441207. No abstract available. PMID 11259725
- [Background] Cohen S, Janicki-Deverts D, Miller GE. Psychological stress and disease. JAMA. 2007 Oct 10;298(14):1685-7. doi: 10.1001/jama.298.14.1685. No abstract available. PMID 17925521
- [Background] DellaGioia N, Hannestad J. A critical review of human endotoxin administration as an experimental paradigm of depression. Neurosci Biobehav Rev. 2010 Jan;34(1):130-43. doi: 10.1016/j.neubiorev.2009.07.014. Epub 2009 Aug 8. PMID 19666048
- [Background] DeRijk RH, Boelen A, Tilders FJ, Berkenbosch F. Induction of plasma interleukin-6 by circulating adrenaline in the rat. Psychoneuroendocrinology. 1994;19(2):155-63. doi: 10.1016/0306-4530(94)90005-1. PMID 8190835
- [Background] Kendler KS, Karkowski LM, Prescott CA. Causal relationship between stressful life events and the onset of major depression. Am J Psychiatry. 1999 Jun;156(6):837-41. doi: 10.1176/ajp.156.6.837. PMID 10360120
- [Background] Kiecolt-Glaser JK, Preacher KJ, MacCallum RC, Atkinson C, Malarkey WB, Glaser R. Chronic stress and age-related increases in the proinflammatory cytokine IL-6. Proc Natl Acad Sci U S A. 2003 Jul 22;100(15):9090-5. doi: 10.1073/pnas.1531903100. Epub 2003 Jul 2. PMID 12840146
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Kleckner IR, Wormwood JB, Simmons WK, Barrett LF, Quigley KS. Methodological recommendations for a heartbeat detection-based measure of interoceptive sensitivity. Psychophysiology. 2015 Nov;52(11):1432-40. doi: 10.1111/psyp.12503. Epub 2015 Aug 12. PMID 26265009
- [Background] Kop WJ, Weissman NJ, Zhu J, Bonsall RW, Doyle M, Stretch MR, Glaes SB, Krantz DS, Gottdiener JS, Tracy RP. Effects of acute mental stress and exercise on inflammatory markers in patients with coronary artery disease and healthy controls. Am J Cardiol. 2008 Mar 15;101(6):767-73. doi: 10.1016/j.amjcard.2007.11.006. Epub 2008 Feb 21. PMID 18328837
- [Background] Miller G, Chen E, Cole SW. Health psychology: developing biologically plausible models linking the social world and physical health. Annu Rev Psychol. 2009;60:501-24. doi: 10.1146/annurev.psych.60.110707.163551. PMID 19035829
- [Background] Nosek, B. A., Banaji, M., & Greenwald, A. G. (2002). Harvesting implicit group attitudes and beliefs from a demonstration web site. Group Dynamics: Theory, Research, and Practice, 6(1), 101-115.
- [Background] Pitman RK, Sanders KM, Zusman RM, Healy AR, Cheema F, Lasko NB, Cahill L, Orr SP. Pilot study of secondary prevention of posttraumatic stress disorder with propranolol. Biol Psychiatry. 2002 Jan 15;51(2):189-92. doi: 10.1016/s0006-3223(01)01279-3. PMID 11822998
- [Background] Raison CL, Miller AH. The evolutionary significance of depression in Pathogen Host Defense (PATHOS-D). Mol Psychiatry. 2013 Jan;18(1):15-37. doi: 10.1038/mp.2012.2. Epub 2012 Jan 31. PMID 22290120
- [Background] Rohleder N. Stimulation of systemic low-grade inflammation by psychosocial stress. Psychosom Med. 2014 Apr;76(3):181-9. doi: 10.1097/PSY.0000000000000049. PMID 24608036
- [Background] Steptoe A, Kivimaki M. Stress and cardiovascular disease. Nat Rev Cardiol. 2012 Apr 3;9(6):360-70. doi: 10.1038/nrcardio.2012.45. PMID 22473079
- [Background] Slavich GM, Irwin MR. From stress to inflammation and major depressive disorder: a social signal transduction theory of depression. Psychol Bull. 2014 May;140(3):774-815. doi: 10.1037/a0035302. Epub 2014 Jan 13. PMID 24417575
- [Background] Slavich GM, Way BM, Eisenberger NI, Taylor SE. Neural sensitivity to social rejection is associated with inflammatory responses to social stress. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14817-22. doi: 10.1073/pnas.1009164107. Epub 2010 Aug 2. PMID 20679216
- [Background] Steptoe A, Hamer M, Chida Y. The effects of acute psychological stress on circulating inflammatory factors in humans: a review and meta-analysis. Brain Behav Immun. 2007 Oct;21(7):901-12. doi: 10.1016/j.bbi.2007.03.011. Epub 2007 May 1. PMID 17475444
- [Background] Emerging Risk Factors Collaboration; Kaptoge S, Di Angelantonio E, Lowe G, Pepys MB, Thompson SG, Collins R, Danesh J. C-reactive protein concentration and risk of coronary heart disease, stroke, and mortality: an individual participant meta-analysis. Lancet. 2010 Jan 9;375(9709):132-40. doi: 10.1016/S0140-6736(09)61717-7. Epub 2009 Dec 22. PMID 20031199
- [Background] Vaiva G, Ducrocq F, Jezequel K, Averland B, Lestavel P, Brunet A, Marmar CR. Immediate treatment with propranolol decreases posttraumatic stress disorder two months after trauma. Biol Psychiatry. 2003 Nov 1;54(9):947-9. doi: 10.1016/s0006-3223(03)00412-8. PMID 14573324
- [Background] van Gool J, van Vugt H, Helle M, Aarden LA. The relation among stress, adrenalin, interleukin 6 and acute phase proteins in the rat. Clin Immunol Immunopathol. 1990 Nov;57(2):200-10. doi: 10.1016/0090-1229(90)90034-n. PMID 1698583
- [Background] Wittenbrink B, Judd CM, Park B. Evidence for racial prejudice at the implicit level and its relationship with questionnaire measures. J Pers Soc Psychol. 1997 Feb;72(2):262-74. doi: 10.1037//0022-3514.72.2.262. PMID 9107001
- [Derived] MacCormack JK, Armstrong-Carter EL, Gaudier-Diaz MM, Meltzer-Brody S, Sloan EK, Lindquist KA, Muscatell KA. beta-Adrenergic Contributions to Emotion and Physiology During an Acute Psychosocial Stressor. Psychosom Med. 2021 Nov-Dec 01;83(9):959-968. doi: 10.1097/PSY.0000000000001009. PMID 34747583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy young adult participants were recruited from campus via flyers and listserv postings. All participants were screened over telephone to ensure they were healthy.
Pre-assignment Details: No enrolled participants were excluded from the study before assignment to groups.
Groups:
- Propanolol Hydrochloride: This is the experimental group given the beta-blocker, propanolol hydrochloride with a single 40mg tablet dosage.
- Placebo: This is the control group given a placebo, which was a single placebo-matching active drug dose.
Period: Overall Study
Arm/Group | Propanolol Hydrochloride | Placebo
Started | 44 | 48
Completed | 44 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propanolol Hydrochloride: This is the experimental group given the beta-blocker, propanolol hydrochloride with a 40mg single tablet dosage.
- Placebo: This is the control group given a placebo, which was a placebo-matching active drug single dosage.
- Total: Total of all reporting groups
Arm/Group | Propanolol Hydrochloride | Placebo | Total
Number analyzed (Participants) | 44 | 48 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 48 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.07 (1.28) | 20.49 (1.56) | 20.28 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 24 | 26 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 25 | 28 | 53
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 48 | 92
Interleukin-6 (IL-6) [Mean (Standard Deviation); unit: log(picograms/mL)] — Measured in blood plasma using enzyme-linked immunosorbent assay. All units are log transformed prior to analysis to correct for skew in data.
  log(picograms/mL) | -1.00 (.90) | -.98 (.86) | -.99 (.88)
Salivary Cortisol [Mean (Standard Deviation); unit: nanomole/L] — Concentration of cortisol in saliva quantified quantified by chemiluminescence immunoassay with high sensitivity.
  nanomole/L | 11.51 (13.04) | 8.62 (12.05) | 10.07 (12.55)
Salivary Alpha-Amylase [Mean (Standard Deviation); unit: picograms/mL] — Concentration of alpha-amylase in saliva quantified by enzyme kinetic method.
  picograms/mL | 44.68 (38.85) | 55.13 (47.17) | 49.91 (43.01)
Pre-Ejection Period [Mean (Standard Deviation); unit: milliseconds] — Derived from impedance cardiography and electrocardiogram.
  milliseconds | 119.97 (18.48) | 116.66 (13.49) | 118.32 (15.99)
Respiratory Sinus Arrhythmia [Mean (Standard Deviation); unit: ratio] — Derived from electrocardiogram; measure of heart rate variability assessed as the ratio of low frequency/high frequency in the respiratory/cardiac power spectrum.
  ratio | 6.86 (1.18) | 7.02 (1.02) | 6.94 (1.10)
Negative, High Arousal Emotion [Mean (Standard Deviation); unit: scores on a scale] — Self-report measure of affect (emotion) state using the Positive and Negative Affect Schedule (PANAS). Answered on a Likert scale from 0 ("not at all") - 6 ("very much"). Mean score range is from 0-6. Higher numbers indicate more negative, high arousal emotions; low numbers indicate less negative, high arousal emotions.
  scores on a scale | 1.20 (.19) | 1.25 (.33) | 1.23 (.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin-6 (IL-6)
Description: Measured in blood plasma using enzyme-linked immunosorbent assay. Log-transformed prior to analysis to correct for skew in data. Four different change scores were calculated: first, change at post-drug from pre-drug baseline; second, the change at 30-min post-stressor from post-drug baseline; third, change at 60-min post-stressor from post-drug baseline; and fourth, change at 90-min post-stressor from post-drug baseline.
Time Frame: Pre-drug baseline; 60-min post-drug administration baseline before stressor; 30-min post-stressor; 60-min post-stressor; 90-min post-stressor
Measure: Mean (95% Confidence Interval); unit: log(picograms/mL)
Groups:
- Propanolol Hydrochloride: This is the experimental group given the beta-blocker, propanolol hydrochloride using a 40mg single tablet dosage.
- Placebo: This is the control group given a placebo, which was a placebo-matching active drug
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
log(picograms/mL)
  Post-drug from pre-drug baseline | .05 [-.126 to .226] | .16 [-.075 to .395]
  30-min post-stress from post-drug baseline | .31 [.016 to .604] | .24 [.044 to .436]
  60-min post-stress from post-drug baseline | .32 [.006 to .634] | .19 [.014 to .366]
  90-min post-stress from post-drug baseline | .48 [.206 to .754] | .46 [.264 to .656]

2. Secondary Outcome: Change in Salivary Cortisol
Description: Concentration of cortisol in saliva quantified quantified by chemiluminescence immunoassay with high sensitivity. Three different change scores were calculated from pre-drug to post-drug baselines, 15-min post-stressor from post-drug baseline, and 30-min post-stressor from post-drug baseline.
Time Frame: Pre-drug baseline; 60-min post-drug administration baseline before stressor; 15-min post-stressor; 30-min post-stressor
Measure: Mean (95% Confidence Interval); unit: nanomole/L
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
nanomole/L
  Post-drug from pre-drug baseline | -6.42 [-8.576 to -4.264] | -3.76 [-5.524 to -1.996]
  15-min post-stress from post-drug baseline | 5.61 [3.258 to 7.962] | 4.02 [2.785 to 5.255]
  30-min post-stress from post-drug baseline | 2.1 [.179 to 4.021] | 1.86 [.978 to 2.742]

3. Secondary Outcome: Change in Salivary Alpha Amylase
Description: Concentration of alpha amylase in saliva quantified quantified by enzyme kinetic method. Two different change scores were calculated: first, the pre-drug to post-drug baseline change and, second, the 15-min post-stressor change from post-drug baseline.
Time Frame: Pre-drug baseline; 60-min post-drug administration baseline before stressor; 15-min post-stressor
Measure: Mean (95% Confidence Interval); unit: picograms / mL
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
picograms / mL
  Post-drug from pre-drug baseline | -7.50 [-19.299 to 4.299] | -6.36 [-16.787 to 4.067]
  15-min post-stress from post-drug baseline | -15.68 [-26.725 to -4.635] | 6.73 [-3.305 to 16.765]

4. Secondary Outcome: Change in Pre-Ejection Period
Description: Mean level pre-ejection period (PEP; centered at zero) derived from impedance cardiography and electrocardiogram. Four different change scores were calculated: first, the change in average PEP from the 5-min pre-drug baseline to the 5-min post-drug baselines; second, the change in average PEP that occurred during the 2-min anticipatory stress speech preparation phase of the Trier Social Stress Test (TSST) from the post-drug baseline; third, the change in average PEP that occurred across the 15-min of the TSST (speech + math tasks) from the post-drug baseline; fourth and finally, the change in average PEP that occurred across 7-min in a post-stressor recovery period as compared to the post-drug baseline.
Time Frame: Pre-drug baseline; 60-min post-drug administration baseline before stressor; 2-min before the stressor; 15-min during stressor, 7-min recovery post-stressor
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
milliseconds
  Post-drug from pre-drug baseline | 7.14 [1.711 to 12.569] | .86 [-3.148 to 4.868]
  TSST-prep from post-drug baseline | -5.33 [-9.828 to -.832] | -10.92 [-14.859 to -6.980]
  TSST from post-drug baseline | -.80 [-6.259 to 4.659] | -10.69 [-14.816 to -6.564]
  Post-stress recovery from post-drug baseline | .21 [-4.063 to 4.483] | -1.19 [-5.120 to 2.740]

5. Secondary Outcome: Change in Respiratory Sinus Arrhythmia
Description: Mean level respiratory sinus arrhythmia (RSA) derived from electrocardiogram; measure of heart rate variability assessed as the ratio of low-to-high frequencies in the respiratory-cardiac power spectrum. Four different change scores were calculated: first, the change in average RSA from the 5-min pre-drug baseline to the 5-min post-drug baselines; second, the change in average RSA that occurred during the 2-min anticipatory stress speech preparation phase of the Trier Social Stress Test (TSST) from the post-drug baseline; third, the change in average RSA that occurred across the 15-min of the TSST (speech + math tasks) from the post-drug baseline; fourth and finally, the change in average RSA that occurred across 7-min in a post-stressor recovery period as compared to the post-drug baseline.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
Ratio
  Post-drug from pre-drug baseline | .11 [-.173 to .395] | .27 [-.025 to .563]
  TSST-prep from post-drug baseline | .36 [.076 to .644] | -.43 [-.734 to -.126]
  TSST from post-drug baseline | -.06 [-.332 to .212] | -.87 [-1.20 to -.540]
  Post-stress recovery from post-drug baseline | .36 [.088 to .632] | -.26 [-.593 to .073]

6. Secondary Outcome: Change in Negative, High Arousal Emotion
Description: Self-report measure of affect (emotion) state using the Positive & Negative Affect Schedule Negative Affect (PANAS). Answered on a Likert scale from 0 ("not at all") - 6 ("very much"). Mean score range is from 0-6. Higher numbers indicate more negative, high arousal emotions; low numbers indicate less negative, high arousal emotions. Three change scores were calculated from the four different rating measurement time points: a change in negative, high arousal emotions at the post-drug baseline from the pre-drug baseline; a change in emotions right before the Trier Social Stress Task (TSST) from the post-drug baseline; and a change in emotions during the TSST from the post-drug baseline.
Time Frame: Pre-drug baseline; 60-min post-drug administration baseline before stressor; 2-min before the stressor; 1-min post-stressor
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propanolol Hydrochloride | Placebo
Number analyzed (Participants) | 44 | 48
score on a scale
  Post-drug from pre-drug baseline | -.10 [-.141 to -.059] | -.13 [-.185 to -.075]
  TSST-prep from post-drug baseline | .18 [.122 to .238] | .37 [.300 to .440]
  TSST stressor from post-drug baseline | .61 [.532 to .689] | .76 [.678 to .842]

ADVERSE EVENTS:
Time Frame: From the time of randomization until 9 months following.
Description: All participants were carefully prescreened to ensure no contra-indications for the low dose (40 mg) of propranolol.
Groups:
- Propanolol Hydrochloride: This is the experimental group given the beta-blocker propanolol hydrochloride. All subjects in this group received a single dose of 40mg of propanolol in a single tablet.
- Placebo: This is the control group given a placebo. All subjects in this group received a single dose of the placebo in a single tablet.
Arm/Group | Propanolol Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/48
Other Adverse Events (participants affected / at risk) | 0/44 | 0/48

LIMITATIONS AND CAVEATS:
1. Not all salivary alpha amylase samples were assayed in duplicate because there was not enough saliva for the 15-min post-stress time point. 2. For the first ten subjects, a shorter version of the PANAS with 20 rather than full 40 items was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT02972554/Prot_SAP_000.pdf